CLINICAL TRIAL: NCT06956872
Title: Clinical Effectiveness of MyNutriKidney® for Dietary Self-management in Chronic Kidney Disease Patients: Protocol for a Pragmatic Randomized Controlled Trial
Brief Title: Clinical Effectiveness of MyNutriKidney®
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: International Society of Nephrology (Other)
Responsible Party: Principal Investigator, Kent Leong Sim Kian, Principle Investigator [Dietitian], Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMRR-19-3569-50972A
Record Dates: First submitted 2025-04-23; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Kidney Disease Stage 3; Chronic Kidney Disease; Chronic Kidney Disease Stage 5; Chronic Kidney Disease Stage 4
Keywords: MyNutriKidney; chronic kidney disease; CKD; Dietary Adherence; Nutrition Literacy; Self-management; Mobile Health; Dietitian; mHealth; Telemedicine; Digital Health; Malaysia; Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care + Renal Diet App (Experimental): Participants receive usual standard care for CKD stages 3-5, supplemented with the use of the MyNutriKidney® mobile application for a 6-month period. Following onboarding and training, participants utilize the app for daily manual meal logging, receive automated nutrient estimations and real-time feedback against personalized dietary recommendations (utilizing a Malaysian food database), access tailored educational modules, engage with gamification features (challenges, progress tracking), and receive periodic personalized feedback from study dietitians via in-app messaging or virtual consultations. Technical support is available.
  Interventions: Other: Counseling; Other: Renal Diet App
- Standard Care (Placebo Comparator): Participants receive usual standard care for CKD stages 3-5 as provided at the participating clinics for a 6-month period. This typically includes face-to-face dietary counseling sessions with a clinic dietitian scheduled based on clinical need (e.g., every 1-3 months), provision of standard printed educational materials and general CKD dietary guidelines, and routine clinical and laboratory monitoring by their usual healthcare providers. Participants in this group do not receive access to the MyNutriKidney® app during the study.
  Interventions: Other: Counseling; Other: Printed Nutrition Pamphlet

INTERVENTIONS:
Other: Counseling — Subjects in the both arms will receive individualized dietetic counseling as the standard dietetic care in Malaysia
Other: Renal Diet App — Individualized dietetic counseling aided with a newly developed renal diet app for educative purpose and aiding tool to enhance the dietary adherence among CKD patients. Training on the use of the app will be provided to the subjects prior to the commencement of the intervention. Subjects will be trained on the use of the home screen, icons, feedback screens, the process of entering dietary and fluid intake data and selecting portion sizes. Subjects are considered as competent users when they could correctly record the foods and drinks with correct portion size eaten in the past 24 hours and successfully save the data.
  Other Names: MyNutriKidney
  Arms: Standard Care + Renal Diet App
Other: Printed Nutrition Pamphlet — After the counseling session, a standardized renal nutrition pamphlet prepared by dietitians from Universiti Putra Malaysia and Hospital Serdang will be given for patient's educative purpose. Since the mobile application is intended for patient's education and self-monitoring (food diary) purposes, and thus, to ensure the comparability between intervention and control groups, the patients in control group will be trained to record their diet intakes manually using the recommended approach 3-day diet records. Nutritional feedback or advices on the diet records will be given to the participants during follow up sessions.
  Arms: Standard Care

SUMMARY:
This study is a 6-month, pragmatic, multi-center, sequentially recruited, stratified, open-label randomized controlled trial (RCT) conducted in Malaysia. It aims to determine the clinical effectiveness of a culturally adapted, gamified mobile health app (MyNutriKidney®) supplementing standard care, compared to standard care alone, for improving dietary self-management among 200 adults with Chronic Kidney Disease (CKD) stages 3-5. Participants will be randomly assigned (1:1, stratified by age and education) into either (i) the intervention group (MyNutriKidney® app + standard care) or (ii) the control group (standard care, including routine dietary counseling and printed materials). The co-primary outcomes are changes in Dietary Adherence (measured by CKD Diet Score) and Nutrition Literacy (measured by NLS score) from baseline to 6 months.

DETAILED DESCRIPTION:
General Objective:

To evaluate the clinical effectiveness of supplementing standard care with the MyNutriKidney® mobile application compared to standard care alone in improving dietary adherence and nutrition literacy among patients with Chronic Kidney Disease (CKD) stages 3-5 in Malaysia over a 6-month period.

Specific Objectives:

1. To compare the change in Dietary Adherence (DA), assessed by the CKD Diet Score (derived from 3x 24-hour dietary recalls), from baseline to 6 months between the MyNutriKidney® intervention group and the standard care control group. (Co-primary objective)
2. To compare the change in Nutrition Literacy (NL), assessed by the Nutrition Literacy Scale (NLS) score, from baseline to 6 months between the intervention and control groups. (Co-primary objective)
3. To compare the changes in secondary outcomes from baseline to 6 months between the two groups, including:

   3.1. Dietary Knowledge, assessed by the Dietary Knowledge Questionnaire (DKQ) score.

   3.2. Kidney Function, assessed by the estimated Glomerular Filtration Rate (eGFR).

   3.3. Serum Electrolyte Levels (Potassium, Phosphorus, Sodium, Calcium).
4. To evaluate app engagement metrics (e.g., meal logging frequency, time spent on educational resources, challenge completion) among participants in the MyNutriKidney® intervention group over the 6-month period. (Exploratory objective)
5. To assess participant satisfaction and usability of the MyNutriKidney® app using the Malay version of the mHealth Application Usability Questionnaire (M-MAUQ) at 6 months among participants in the intervention group. (Exploratory objective)

ELIGIBILITY:
Participants must meet all of the following inclusion criteria and none of the exclusion criteria to be eligible for enrolment into the study.

Inclusion Criteria:

1. Clinically diagnosed Chronic Kidney Disease (CKD):

   1.1. eGFR < 60 ml/min/1.73m² for ≥ 3 months (applicable to pre-dialysis patients, Stages 3-5)
2. Aged 18 years or older.
3. Possesses a personal smartphone compatible with the MyNutriKidney® application and is willing to use the health app if randomized to the intervention group.
4. Alert and oriented, and deemed capable of providing informed consent and participating in study procedures.
5. Able to communicate and understand study procedures in English, Bahasa Melayu, or Mandarin.

Exclusion Criteria:

1. Inability to effectively use the smartphone application due to significant impairments (e.g., severe visual or motor problems).
2. Smartphone owned by the participant does not meet the minimum technical requirements for the MyNutriKidney® application installation and operation
3. Presence of significant cognitive impairment or severe psychological conditions (e.g., uncontrolled anxiety or depression) likely to impede consistent participation or adherence to study requirements.
4. Known unwillingness or inability to comply with core study procedures, including dietary assessment components.
5. Concurrent participation in another interventional research study.
6. Participation in another research study involving an investigational product in the 12 weeks preceding potential enrollment.
7. Female participants who are pregnant, currently lactating, or planning a pregnancy during the course of the trial.
8. Currently receiving primary nutritional support via enteral tube feeding or parenteral (intra-venous) nutrition.
9. Currently receiving active treatment for cancer (e.g., chemotherapy, radiotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary Adherence Score | Change from Baseline (Month 0) to 6 Months (Month 6).
  Dietary Adherence (DA) quantified using CKD Diet Score (adapted from GCKD study). Intake data from 3x 24-hour dietary recalls (dietitian interview) per assessment (Baseline, M3, M6). Nutrient intake analyzed.
  Score derived from 6 components: sodium, potassium, fiber, total protein, sugar, cholesterol. Intake adjusted per 1000 kcal; points 1 (poor) to 5 (high adherence) assigned based on thresholds.
  Sodium and total protein scores weighted x1.5. Total Score = (Sodium Score 1.5) + Potassium Score + Fiber Score + (Protein Score 1.5) + Sugar Score + Cholesterol Score.
  Total score range: 7 (poorest adherence) to 35 (highest adherence).
Change in Nutrition Literacy Score | Change from Baseline (Month 0) to 6 Months (Month 6).
  Nutrition Literacy assessed using the Nutrition Literacy Scale (NLS) score (validated Malay version). The standardized index score ranges from 0 (lowest literacy) to 100 (highest literacy).

SECONDARY OUTCOMES:
Change in Dietary Knowledge Score | Change from Baseline (Month 0) to 6 Months (Month 6).
  Dietary Knowledge assessed using the Dietary Knowledge Questionnaire (DKQ) score (25 items). Score is expressed as a percentage (0-100%), with higher scores indicating greater knowledge
Change in Estimated Glomerular Filtration Rate (eGFR) | Change from Baseline (Month 0) to 6 Months (Month 6)
  eGFR calculated using the CKD-EPI formula based on serum creatinine levels extracted from routine clinical laboratory results. Measured in mL/min/1.73 m².
Change in Serum Albumin Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Serum Albumin level extracted from routine clinical laboratory results. Units measured according to local laboratory standards (e.g., g/L).
Change in Hemoglobin Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Hemoglobin level extracted from routine clinical laboratory results. Units measured according to local laboratory standards (e.g., g/dL).
Change in Serum Potassium Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Serum potassium (K) level extracted from routine clinical laboratory results obtained near the study visit time points as part of standard CKD care. Unit: mmol/L.
Change in Serum Phosphorus Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Serum phosphorus (P) level extracted from routine clinical laboratory results obtained near the study visit time points as part of standard CKD care. Unit: mmol/L.
Change in Serum Sodium Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Serum sodium (Na) level extracted from routine clinical laboratory results obtained near the study visit time points as part of standard CKD care. Unit: mmol/L.
Change in Corrected Serum Calcium Level | Change from Baseline (Month 0) to 6 Months (Month 6).
  Corrected serum calcium (Ca) level extracted from routine clinical laboratory results obtained near the study visit time points as part of standard CKD care. Unit: mmol/L.

OTHER OUTCOMES:
App Usability and Satisfaction Score | Assessed at 6 Months (Month 6).
  Assessed using the Malay version of the mHealth Application Usability Questionnaire (M-MAUQ). An overall average score is calculated based on a 7-point Likert scale (1=strongly disagree to 7=strongly agree), with higher scores indicating better usability/satisfaction. (Assessed in Intervention Group only).
Average Weekly Meal Logging Frequency | Calculated as an average over the period from Baseline (Month 0) to 6 Months (Month 6).
  Frequency of meal logging, calculated as average logs per week, derived from passively logged user interaction data from the MyNutriKidney® app's backend analytics system. Unit: logs/week. (Assessed in Intervention Group only).
Average Weekly Time on Educational Modules | Calculated as an average over the period from Baseline (Month 0) to 6 Months (Month 6).
  Time spent interacting with educational modules, calculated as average minutes per week, derived from passively logged user interaction data from the MyNutriKidney® app's backend analytics system. Unit: minutes/week. (Assessed in Intervention Group only).
Total Number of Gamification Challenges Completed | Calculated as a total over the period from Baseline (Month 0) to 6 Months (Month 6).
  Completion of gamification challenges, measured as the total number completed, derived from passively logged user interaction data from the MyNutriKidney® app's backend analytics system. Unit: count. (Assessed in Intervention Group only).
Interaction Rate with Actionable Reminders | Calculated over the period from Baseline (Month 0) to 6 Months (Month 6)
  Responsiveness to notifications, measured as the interaction rate with actionable reminders, derived from passively logged user interaction data from the MyNutriKidney® app's backend analytics system. (Number of Interactions / Number of Reminders Sent) * 100%. Unit: %. (Assessed in Intervention Group only).

CONTACTS AND LOCATIONS:
Overall Officials: Nor Fadhlina binti Zakaria, Nephrologist, Principal Investigator — Universiti Putra Malaysia; Barakatun Nisak binti Mohd Yusof, Dietitian Professor [Dr], Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Sultan Idris Shah Hospital, Serdang, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saminathan TA, Hooi LS, Mohd Yusoff MF, Ong LM, Bavanandan S, Rodzlan Hasani WS, Tan EZZ, Wong I, Rifin HM, Robert TG, Ismail H, Wong NI, Ahmad G, Ambak R, Othman F, Abd Hamid HA, Aris T. Prevalence of chronic kidney disease and its associated factors in Malaysia; findings from a nationwide population-based cross-sectional study. BMC Nephrol. 2020 Aug 14;21(1):344. doi: 10.1186/s12882-020-01966-8. PMID 32795256
- [Background] Campbell J, Porter J. Dietary mobile apps and their effect on nutritional indicators in chronic renal disease: A systematic review. Nephrology (Carlton). 2015 Oct;20(10):744-751. doi: 10.1111/nep.12500. PMID 25959301
- [Background] Lim JH, Lim CK, Ibrahim I, Syahrul J, Mohamed Zabil MH, Zakaria NF, Daud ZAM. Limitations of Existing Dialysis Diet Apps in Promoting User Engagement and Patient Self-Management: Quantitative Content Analysis Study. JMIR Mhealth Uhealth. 2020 Jun 1;8(6):e13808. doi: 10.2196/13808. PMID 32478665
- [Background] Lim JH, Chinna K, Khosla P, Karupaiah T, Daud ZAM. Understanding How Nutrition Literacy Links to Dietary Adherence in Patients Undergoing Maintenance Hemodialysis: A Theoretical Exploration Using Partial Least Squares Structural Equation Modeling. Int J Environ Res Public Health. 2020 Oct 14;17(20):7479. doi: 10.3390/ijerph17207479. PMID 33066603
- [Background] Thong KM, Jalalonmuhali M, Choo CL, Yee SY, Yahya R, Jeremiah PN, Bavanandan S, Hooi LS. Audit on data accuracy of the Malaysian Dialysis and Transplant Registry (MDTR). Med J Malaysia. 2024 Mar;79(2):234-236. PMID 38553931